CLINICAL TRIAL: NCT02385006
Title: Thromboelastographic Profile During Simultaneous Pancreas-kidney Transplantation
Brief Title: Thromboelastography and Pancreas-kidney Transplantation
Acronym: TEG-PKT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2012.727
Record Dates: First submitted 2015-02-26; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Blood Coagulation
Keywords: Thromboelastography; simulatneous pancreas-kidney transplantation
MeSH Terms: conditions — Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm kidney transplanted (Other): Arm kidney transplanted: all patients who receive kidney transplantation
  Interventions: Biological: Blood sample
- Arm pancreas-kidney transplanted (Other): Arm pancreas-kidney transplanted: all patients who receive pancreas-kidney transplantation
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample

SUMMARY:
Type of study:Prospective, single-center, non-therapeutic, of routine care No randomization, no modifications of the usual care, study results are not available for the physicians in charge of the patient.

Objectives:

* The main objective of this study is to evaluate the ability of the thromboelastogram (ROTEM®) to detect clotting disorders related to pancreas-kidney transplantation, comparing ROTEM ® profiles during the perioperative period of two different types of transplantation (kidney alone and simultaneous pancreas-kidney)
* The secondary objectives are:

  1. To assess the incidence and type of coagulation disorders during the perioperative period of these two types of transplantation
  2. To study correlation values between thrombolelastogram and standard coagulation parameters

Population study:

* Evaluated group: 40 pancreas-kidney recipients
* Control group: 80 kidney recipients
* Recruitment periods: 24 months
* Patient Monitoring: 48 hours
* Total duration of the study: 36 months.
* Ethics: Study of routine care. Oral and written information given to patients. Validation of the study protocol by the local ethics committee (CPP Sud Est II: Protocol No. HCL / P 2012.727)

ELIGIBILITY:
Inclusion Criteria:

* Men, women > 18 years old
* Kidney or pancreas-kidney recipients
* Not opposed to research
* With no legal protection
* Affiliated to social security system

Exclusion Criteria:

-Enrollment in an other research protocol, incompatible with the trial according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Thromboelastogram (ROTEM®) channels (APTEM, EXTEM, INTEM, FIBTEM) monitoring | preoperative period
Thromboelastogram (ROTEM®) channels (APTEM, EXTEM, INTEM, FIBTEM) monitoring | 45 min after transplant unclamp
Thromboelastogram (ROTEM®) channels (APTEM, EXTEM, INTEM, FIBTEM) monitoring | Intensice Care Unit admission
Thromboelastogram (ROTEM®) channels (APTEM, EXTEM, INTEM, FIBTEM) monitoring | 24 hours
Thromboelastogram (ROTEM®) channels (APTEM, EXTEM, INTEM, FIBTEM) monitoring | 48 hours

SECONDARY OUTCOMES:
standard coagulation parameters | preoperative period
standard coagulation parameters | 45 min after transplant unclamp
standard coagulation parameters | Intensice Care Unit admission
standard coagulation parameters | 24 hours
standard coagulation parameters | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Critical Care Medicine, Edouard Herriot Hospital, Hospices Civils de Lyon, Lyon, France